CLINICAL TRIAL: NCT04479501
Title: Retrospective Review on Patients With Recurrent Asthmatic Attacks Requiring Hospitalizations
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: United Christian Hospital (Other); Princess Margaret Hospital, Hong Kong (Other Government); Pamela Youde Nethersole Eastern Hospital (Other); Queen Elizabeth Hospital, Hong Kong (Other); Queen Mary Hospital, Hong Kong (Other); Kwong Wah Hospital (Other); Tseung Kwan O Hospital, Hong Kong (Other); Caritas Medical Centre, Hong Kong (Other); North District Hospital, Hong Kong (Unknown); Alice Ho Miu Ling Nethersole Hospital (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Honorary Clinical Tutor, Chinese University of Hong Kong
Other Study IDs: CREC 2017.503
Record Dates: First submitted 2020-06-28; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Asthma; Asthma exacerbation; Asthma hospitalization; Asthma control; Asthma care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma group: Patients with asthma
  Interventions: Other: Asthma exacerbation related hospitalization

INTERVENTIONS:
Other: Asthma exacerbation related hospitalization — Evaluate the difference between patients with single and multiple hospitalizations for asthma exacerbation

SUMMARY:
Asthma is a common respiratory disease. around the world. Asthma exacerbation is one of the major sequelae and associated with various morbidity and mortality. A satisfactory asthma control can help to bring down the risk of exacerbation and hence hospitalization. However, the real-world evidence on the clinical factors that leads to multiple admissions, when compared with single admission, due to asthma exacerbation is scarce. This study aimed at evaluating the clinical characteristics of patients who had single and multiple hospitalizations for asthma exacerbations, and exploring the risk factors that predict multiple hospitalizations.

DETAILED DESCRIPTION:
Asthma is a common respiratory disease worldwide and in Hong Kong. According to the estimation by the Center for Disease Control and Prevention in 2015, 7.6% adults in the United States have asthma. In Hong Kong, the prevalence of asthma was estimated to be 10.1% among 13 to 14 years old children and 5.8% in randomly selected Chinese elderly aged more than 70. The clinical characteristics varies in different age groups, with elderly asthmatics have higher rates of bronchial hyper-reactivity and more severe phenotypes, when comparing with younger patients. This is more important in an ageing population.

Asthmatic exacerbation is not an uncommon complication and can be fatal. For those patients with near-fatal asthma exacerbation, ICU admission and mechanical ventilation may be necessary to prevent mortality. This is more common among poor controllers and adults. Asthma-related deaths may be reduced if risk factors are recognized and addressed early.

Many predictors for exacerbation had been identified, both endogenous and exogenous, including high eosinophil count, upper airway diseases, gastroesophageal reflux, poor inhaler technique, medication non-compliance, guideline non-compliance. One of the most powerful predictors for future exacerbation in patients with severe or difficult-to-treat asthma is a recent severe asthma exacerbation. In addition, hospitalization for exacerbations requiring ICU care and mechanical ventilation are both predictors for near-fatal asthma. After the acute attack, its unfavourable impact continues and can lead to multiple sequelae. Exacerbation of asthma is associated with a more rapid decline in the post-bronchodilator forced expiratory volume in 1 second and worse quality of life. In addition, individuals with uncontrolled asthma had higher medical expenditures and decreased productivity, contributing to a greater economic burden when compared with individuals without asthma. In contrary, patients with controlled asthma had lower hospitalization rate, mortality rate and less decline in lung function.

Many of these factors are potentially reversible. But, there is still a significant proportion of asthma patients experiencing recurrent exacerbation despite optimization of pharmacological treatment. A model of better asthma care may be established by improving the understanding on these risk factors, leading to less exacerbation events.

ELIGIBILITY:
Inclusion Criteria:

* All patients with hospitalization for asthmatic exacerbation according to physician's clinical judgement
* Age greater than 18 years old

Exclusion Criteria:

- Inappropriate diagnosis of asthma exacerbation after evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: By using the International Classification of Diseases, Ninth Revision, Clinical Modification code 493.xx, each participating hospital identified all primary hospital discharge diagnosis of asthma (exacerbation) during a 12-month period, between 1st January 2016 to 31st December 2016
Sampling Method: Non-Probability Sample
Enrollment: 2280 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who had hospitalization for asthma attack | 1 year
  Number of patients who had hospitalization for asthma attack

SECONDARY OUTCOMES:
Burden of comorbidity among subjects with recurrent hospital admission for asthma attack | 1 year
  Burden of comorbidity among subjects with recurrent hospital admission for asthma attack
Spirometric parameters (FEV1, FVC) among subjects with recurrent hospital admission for asthma attack | 1 year
  Spirometric parameters (FEV1, FVC) among subjects with recurrent hospital admission for asthma attack
Baseline blood eosinophil among subjects with recurrent hospital admission for asthma attack | 1 year
  Baseline blood eosinophil among subjects with recurrent hospital admission for asthma attack
Prevalence of asthma patients who had received phenotypic workup | 1 year
  Prevalence of asthma patients who had received phenotypic workup

CONTACTS AND LOCATIONS:
Overall Officials: Ka Pang Chan, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: upon individual approach for metaanalysis or related study

REFERENCES:
- [Background] Wong GW, Leung TF, Ko FW. Changing prevalence of allergic diseases in the Asia-pacific region. Allergy Asthma Immunol Res. 2013 Sep;5(5):251-7. doi: 10.4168/aair.2013.5.5.251. Epub 2013 Mar 18. PMID 24003381
- [Background] Ko FW, Lai CK, Woo J, Ho SC, Ho CW, Goggins W, Hui DS. 12-year change in prevalence of respiratory symptoms in elderly Chinese living in Hong Kong. Respir Med. 2006 Sep;100(9):1598-607. doi: 10.1016/j.rmed.2005.12.007. Epub 2006 Jan 30. PMID 16446081
- [Background] Pasha MA, Sundquist B, Townley R. Asthma pathogenesis, diagnosis, and management in the elderly. Allergy Asthma Proc. 2017 May 1;38(3):184-191. doi: 10.2500/aap.2017.38.4048. PMID 28441988
- [Background] Romagnoli M, Caramori G, Braccioni F, Ravenna F, Barreiro E, Siafakas NM, Vignola AM, Chanez P, Fabbri LM, Papi A; ENFUMOSA Study Group. Near-fatal asthma phenotype in the ENFUMOSA Cohort. Clin Exp Allergy. 2007 Apr;37(4):552-7. doi: 10.1111/j.1365-2222.2007.02683.x. PMID 17430352
- [Background] Miller MK, Lee JH, Miller DP, Wenzel SE; TENOR Study Group. Recent asthma exacerbations: a key predictor of future exacerbations. Respir Med. 2007 Mar;101(3):481-9. doi: 10.1016/j.rmed.2006.07.005. Epub 2006 Aug 17. PMID 16914299
- [Background] Dougherty RH, Fahy JV. Acute exacerbations of asthma: epidemiology, biology and the exacerbation-prone phenotype. Clin Exp Allergy. 2009 Feb;39(2):193-202. doi: 10.1111/j.1365-2222.2008.03157.x. PMID 19187331
- [Background] Zeiger RS, Schatz M, Dalal AA, Chen W, Sadikova E, Suruki RY, Kawatkar AA, Qian L. Blood Eosinophil Count and Outcomes in Severe Uncontrolled Asthma: A Prospective Study. J Allergy Clin Immunol Pract. 2017 Jan-Feb;5(1):144-153.e8. doi: 10.1016/j.jaip.2016.07.015. Epub 2016 Sep 21. PMID 27665383
- [Background] Price DB, Rigazio A, Campbell JD, Bleecker ER, Corrigan CJ, Thomas M, Wenzel SE, Wilson AM, Small MB, Gopalan G, Ashton VL, Burden A, Hillyer EV, Kerkhof M, Pavord ID. Blood eosinophil count and prospective annual asthma disease burden: a UK cohort study. Lancet Respir Med. 2015 Nov;3(11):849-58. doi: 10.1016/S2213-2600(15)00367-7. Epub 2015 Oct 19. PMID 26493938
- [Background] ten Brinke A, Sterk PJ, Masclee AA, Spinhoven P, Schmidt JT, Zwinderman AH, Rabe KF, Bel EH. Risk factors of frequent exacerbations in difficult-to-treat asthma. Eur Respir J. 2005 Nov;26(5):812-8. doi: 10.1183/09031936.05.00037905. PMID 16264041
- [Background] Engelkes M, Janssens HM, de Jongste JC, Sturkenboom MC, Verhamme KM. Medication adherence and the risk of severe asthma exacerbations: a systematic review. Eur Respir J. 2015 Feb;45(2):396-407. doi: 10.1183/09031936.00075614. Epub 2014 Oct 16. PMID 25323234
- [Background] Nestor A, Calhoun AC, Dickson M, Kalik CA. Cross-sectional analysis of the relationship between national guideline recommended asthma drug therapy and emergency/hospital use within a managed care population. Ann Allergy Asthma Immunol. 1998 Oct;81(4):327-30. doi: 10.1016/S1081-1206(10)63124-9. PMID 9809496
- [Background] Williams LK, Peterson EL, Wells K, Ahmedani BK, Kumar R, Burchard EG, Chowdhry VK, Favro D, Lanfear DE, Pladevall M. Quantifying the proportion of severe asthma exacerbations attributable to inhaled corticosteroid nonadherence. J Allergy Clin Immunol. 2011 Dec;128(6):1185-1191.e2. doi: 10.1016/j.jaci.2011.09.011. Epub 2011 Oct 21. PMID 22019090
- [Background] Hasegawa K, Sullivan AF, Tovar Hirashima E, Gaeta TJ, Fee C, Turner SJ, Massaro S, Camargo CA Jr; Multicenter Airway Research Collaboration-36 Investigators. A multicenter observational study of US adults with acute asthma: who are the frequent users of the emergency department? J Allergy Clin Immunol Pract. 2014 Nov-Dec;2(6):733-40. doi: 10.1016/j.jaip.2014.06.012. Epub 2014 Sep 10. PMID 25439365
- [Background] Serrano-Pariente J, Plaza V. Near-fatal asthma: a heterogeneous clinical entity. Curr Opin Allergy Clin Immunol. 2017 Feb;17(1):28-35. doi: 10.1097/ACI.0000000000000333. PMID 27870665
- [Background] Turner MO, Noertjojo K, Vedal S, Bai T, Crump S, Fitzgerald JM. Risk factors for near-fatal asthma. A case-control study in hospitalized patients with asthma. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1804-9. doi: 10.1164/ajrccm.157.6.9708092. PMID 9620909
- [Background] Bai TR, Vonk JM, Postma DS, Boezen HM. Severe exacerbations predict excess lung function decline in asthma. Eur Respir J. 2007 Sep;30(3):452-6. doi: 10.1183/09031936.00165106. Epub 2007 May 30. PMID 17537763
- [Background] O'Byrne PM, Pedersen S, Lamm CJ, Tan WC, Busse WW; START Investigators Group. Severe exacerbations and decline in lung function in asthma. Am J Respir Crit Care Med. 2009 Jan 1;179(1):19-24. doi: 10.1164/rccm.200807-1126OC. Epub 2008 Oct 31. PMID 18990678
- [Background] Luskin AT, Chipps BE, Rasouliyan L, Miller DP, Haselkorn T, Dorenbaum A. Impact of asthma exacerbations and asthma triggers on asthma-related quality of life in patients with severe or difficult-to-treat asthma. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):544-52.e1-2. doi: 10.1016/j.jaip.2014.02.011. Epub 2014 Jul 3. PMID 25213047
- [Background] Sullivan PW, Slejko JF, Ghushchyan VH, Sucher B, Globe DR, Lin SL, Globe G. The relationship between asthma, asthma control and economic outcomes in the United States. J Asthma. 2014 Sep;51(7):769-78. doi: 10.3109/02770903.2014.906607. Epub 2014 Apr 7. PMID 24697738
- [Background] Moorman JE, Akinbami LJ, Bailey CM, Zahran HS, King ME, Johnson CA, Liu X. National surveillance of asthma: United States, 2001-2010. Vital Health Stat 3. 2012 Nov;(35):1-58. PMID 24252609
- [Background] Heaney LG, Conway E, Kelly C, Johnston BT, English C, Stevenson M, Gamble J. Predictors of therapy resistant asthma: outcome of a systematic evaluation protocol. Thorax. 2003 Jul;58(7):561-6. doi: 10.1136/thorax.58.7.561. PMID 12832665
- [Background] Robinson DS, Campbell DA, Durham SR, Pfeffer J, Barnes PJ, Chung KF; Asthma and Allergy Research Group of the National Heart and Lung Institute. Systematic assessment of difficult-to-treat asthma. Eur Respir J. 2003 Sep;22(3):478-83. doi: 10.1183/09031936.03.00017003. PMID 14516138
- [Background] Hekking PW, Wener RR, Amelink M, Zwinderman AH, Bouvy ML, Bel EH. The prevalence of severe refractory asthma. J Allergy Clin Immunol. 2015 Apr;135(4):896-902. doi: 10.1016/j.jaci.2014.08.042. Epub 2014 Oct 16. PMID 25441637
- [Background] Koga T, Oshita Y, Kamimura T, Koga H, Aizawa H. Characterisation of patients with frequent exacerbation of asthma. Respir Med. 2006 Feb;100(2):273-8. doi: 10.1016/j.rmed.2005.05.017. Epub 2005 Jul 5. PMID 15998585
- See also: Assessed on 28 April 2017 — http://www.cdc.gov/asthma/most_recent_data.htm